CLINICAL TRIAL: NCT00517842
Title: A Triple-blinded, Randomised, Placebo-controlled Trial to Examine the Efficacy and Safety of ViNeuro in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Vigconic (International) Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2005-228-T; HARECCTR0500017
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Drug: ViNeuro

SUMMARY:
The investigational product is a specially formulated TCM and administered in the form of a capsule.

Basic pre-clinical studies have suggested that it may have good immunomodulating functions, increases the activities of T-cells, B-cells and NK cells, enhances mitochondrial antioxidant status on various tissues including brain tissues. Therefore, this formulation may have special values in improving symptoms in Parkinson's disease patients.

The purpose of the study is to determine the efficacy and safety of ViNeuro in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for study participation if he/she meets all the following criteria:

  1. Age of at least 30 years
  2. Diagnosis of symptomatic, idiopathic Parkinson' disease using The United Kingdom Parkinson's Disease Society Brain Bank Diagnostic Criteria (Appendix 3 in the protocol)
  3. Stage 1-4 on the modified Hoehn and Yahr scale (Appendix 4 in the protocol)
  4. Possesses three of the four cardinal signs of Parkinson's disease, i.e. rigidity, bradykinesia, resting tremor and postural instability, without any other known or suspected cause for their parkinsonism
  5. If receiving levodopa or other symptomatic treatments, the subject should have shown a good response to it and have been on a stable dosage for at least 1 month prior to study entry
  6. Voluntarily signs and dates an Informed Consent Form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to any study-specific procedures.

Exclusion Criteria:

* A subject will be excluded from the study if he/she meets any of the following criteria:

  1. Presence of atypical parkinsonian syndromes
  2. Dementia as defined by the Mini-Mental State Examination score (Appendix 5 in the protocol) of 22 or less
  3. Serious concurrent illness, such as active cardiac, renal, liver, or neoplastic disease
  4. Used centrally active therapies, e.g. hypnotics, antidepressants, anxiolytics, within 60 days before study entry
  5. Used methylphenidate, cinnarizine, reserpine, amphetamine, or monoamine oxidase-A inhibitors, e.g. pargyline, phenelzine, or tranylcpromine, within 3 months of study entry
  6. Has history of receiving any neuroleptics
  7. Used alpha-methyldopa or flunarizine within 6 months of study entry
  8. Females who are pregnant or breastfeeding.
  9. Subjects who are currently participating in another investigational study or has been taking any investigational drug within the last 4 weeks prior to screening of this study (Visit 1).
  10. Subjects who are taking any traditional Chinese medication, or has been taking any traditional Chinese medication within the last 2 weeks prior to screening of this study (Visit 1).
  11. Any criteria, which, in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol.

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2005-10; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome is the change from baseline in the sum of the Unified Parkinson's Disease Rating Scale (UPDRS) (Appendix 6) Parts II and III total scores at the end of 24 weeks. The UPDRS is to be performed one hour after L-dopa treatment. | 24 Weeks

SECONDARY OUTCOMES:
Change from baseline in the individual Part II and Part III total scores, sum of Parts I-III total scores, Part IV total score of the UPDRS at each follow-up visit... | 24 weeks
Change from baseline in the number of "off" hours throughout the study at each follow-up visit. | The mean number of daily "off" hours over the last 7 days before each study visit, except for the screening visit, will be used for the analysis.
Change from baseline in the total daily dose in patients who received concomitant levodopa therapy throughout the study at each follow-up visit; Change from baseline in Red Cell Superoxide Dismutase Activity at 24 week. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonas HM Yeung, Dr, Principal Investigator — Department of Medicine and Therapeutics, Prince of Wales Hospital/ The Chinese University of Hong Kong
Locations (5):
- China (5):
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Tseung Kwan O Hospital, Hong Kong
  - United Christian Hospital, Hong Kong